CLINICAL TRIAL: NCT07028606
Title: Effect of Arginine - Glycine - Aspartic Acid (RGD) Hydrogel on Vertical Ridge Augmentation Using Computer-guided Sandwich Osteotomy Technique, With Xenograft and Simultaneous Implant Placement
Brief Title: Vertical Ridge Augmentation Using Computer-guided Sandwich Osteotomy Technique
Acronym: RGD
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Ahmed Khairy morsi, Assistant Iecturer at Oral Medicine, Periodontology, Oral Radiology and Oral Diagnosis, Faculty of Oral and Dental Medicine, Al-Azhar University, Principal Investigator., Al-Azhar University
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: Arginine - Glycine - Aspartic
Record Dates: First submitted 2025-04-17; First posted 2025-06-19 (Actual); Last update posted 2025-06-19 (Actual); Status verified 2025-06

CONDITIONS: Alveolar Bone Resorption
MeSH Terms: interventions — Transplantation, Heterologous; arginyl-glycyl-aspartic acid

STUDY DESIGN:
Intervention Model Description: The patients will be randomly assigned into two groups; Group 1: (Control group) will receive computer-guided sandwich osteotomy technique with xenograft, collagen membrane and simultaneous implant placement. Group 2: (Study group) will receive computer-guided sandwich osteotomy technique with (RGD), xenograft, collagen membrane and simultaneous implant placement.
Who Masked: Outcomes Assessor
Masking Description: Patients will be randomly assigned to either test or control groups using computer generated randomization (www.randomizer.org)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Sandwich technique with xenograft, collagen membrane and simultaneous implant placement (Placebo Comparator): (Control group) will receive computer-guided sandwich osteotomy technique with xenograft, collagen membrane and simultaneous implant placement.
  Interventions: Procedure: Sandwich technique with xenograft, collagen membrane and simultaneous implant placement.
- Sandwich technique with (RGD), xenograft, collagen membrane and simultaneous implant placement (Active Comparator): (Study group) will receive computer-guided sandwich osteotomy technique with (RGD), xenograft, collagen membrane and simultaneous implant placement.
  Interventions: Biological: Sandwich technique with (RGD), xenograft, collagen membrane and simultaneous implant placement.

INTERVENTIONS:
Procedure: Sandwich technique with xenograft, collagen membrane and simultaneous implant placement. — All surgery will be in upper arch, for sandwich osteotomy technique, after local anesthesia, crestal incision with buccal intrasulcular incisions will be done extending at least one tooth mesial and distal to the implant associated site. Full thickness mucoperiosteal flaps will be reflected to allow access for implant, distraction osteogenesis, xenograft.
  Osteotomy for implant will be carried out with advanced kit of roott_system Switzerland brand, sandwich osteotomy technique will be carried out with three full thickness cuts using the tungsten carbide disc were performed in the form of two vertical cuts away from the neighboring teeth by 3 mm and one horizontal bony cut on the labial surface of alveolar ridge. Bone splitting chisels were used in sequential width (2 mm, 3 mm) and lightweight mallet to complete splitting of the bony segment, the surgical sites will be irrigated with sterile saline. Surgical flaps will be sutured to the pre-surgical level.
  Arms: Sandwich technique with xenograft, collagen membrane and simultaneous implant placement
Biological: Sandwich technique with (RGD), xenograft, collagen membrane and simultaneous implant placement. — All surgery will be in upper arch, for sandwich osteotomy technique, after local anesthesia, crestal incision with buccal intrasulcular incisions will be done extending at least one tooth mesial and distal to the implant associated site. Full thickness mucoperiosteal flaps will be reflected to allow access for implant, distraction osteogenesis, xenograft with and with RGD.
  Injectable RGD-bioconjugate Mussel Adhesive Proteins (RGD-MAPs) composite hydroxypropyl methylcellulose (HPMC) hydrogels . Previously we developed a novel type of injectable self-supported hydrogel (2 mg/ml of RGD-MAPs/HPMC) based porcine nano hydroxyapatite (MPH) for dental graft, which could good handling property, biodegradation or biocompatibility with the hydrogel disassembly and provided efficient cell adhesion activity and no inflammatory responses. Surgical flaps will be sutured to the pre-surgical level with 4-0 polyproline non resorbable suture utilizing a single interrupted suturing technique.
  Arms: Sandwich technique with (RGD), xenograft, collagen membrane and simultaneous implant placement

SUMMARY:
Researcher will introduce the trial to patients and provide full explanation of its aim and benefits in Arabic language. Patients will then be able to have an informed discussion with the researcher. Researcher will obtain written consent from patients willing to participate in the trial

DETAILED DESCRIPTION:
This protocol and the template informed consent form will be reviewed by the Ethics Committee of Scientific Research -Faculty of Oral and Dental Medicine- Al-Azhar University.

ELIGIBILITY:
Inclusion criteria

* Adults (age 30-45) with vertical ridge deficiency.
* Patients with maxillary vertical ridge deficiency 4-8mm according to Cologne Classification of Alveolar Ridge Defects (CCARD).
* Patients with good oral hygiene.
* Free from systemic diseases that may influence the outcome of the therapy.

Exclusion criteria

* Systemic conditions which are generally considered to be a contraindication to implant surgery which included but not limited to: osteoporosis, uncontrolled diabetes.
* Pregnant or lactating females
* Current or former smokers.
* Patient treated by immunosuppressive chemotherapy or radio therapy,
* Allergy to any material or medication used in the study.

Ages: 30 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2024-05-09 (Actual); Primary Completion 2025-05-10 (Actual); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Effect of RGD on volumetric bone changes | Preoperative Cone beam computed tomography (CBCT) with minimal field of view will be taken for (implant treatment plan), immediately after surgery, at time of loading and 6 months after loading.
  Cone beam computed tomography with minimal field of view was taken immediately after surgery, immediately before loading (6 months) and 6 months after loading to evaluate volumetric changes.

CONTACTS AND LOCATIONS:
Locations (1):
- Al-Azhar University, Cairo, Boys, Cairo, Nasr City, Egypt

IPD SHARING:
Plan to Share IPD: No